CLINICAL TRIAL: NCT04472429
Title: A Phase 3 Global, Multicenter, Double-Blind Randomized Study of Carboplatin-Paclitaxel With INCMGA00012 or Placebo in Participants With Inoperable Locally Recurrent or Metastatic Squamous Cell Carcinoma of the Anal Canal Not Previously Treated With Systemic Chemotherapy (POD1UM-303/InterAACT 2)
Brief Title: Carboplatin-paclitaxel With Retifanlimab or Placebo in Participants With Locally Advanced or Metastatic Squamous Cell Anal Carcinoma (POD1UM-303/InterAACT 2).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCMGA 0012-303; 2024-512331-72-00 (Registry Identifier: EU CT Number); 2020-000826-24 (EudraCT Number)
Expanded Access: NCT06910137 (Available)
Record Dates: First submitted 2020-07-13; First posted 2020-07-15 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Squamous Cell Carcinoma of the Anal Canal
Keywords: Squamous cell carcinoma; carboplatin; paclitaxel; PD-1 Inhibitor; Anal Cancer; SCAC
MeSH Terms: conditions — Carcinoma, Squamous Cell; Anus Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A : carboplatin+paclitaxel+placebo (Placebo Comparator): Participants will receive carboplatin on Day 1,paclitaxel on Day1,8, 15, and placebo on Day 1 of each 28 day cycle
  Interventions: Drug: carboplatin; Drug: paclitaxel
- Group B : carboplatin+paclitaxel+retifanlimab (Experimental): Participants will receive carboplatin on Day 1,paclitaxel on Day1,8, 15, and retifanlimab on Day 1 of each 28 day cycle
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: retifanlimab

INTERVENTIONS:
Drug: carboplatin — carboplatin will be administered intravenous on Day 1 of each 28 day cycle
Drug: paclitaxel — paclitaxel will be administered intravenous on Days 1,8, and 15 of each 28 day cycle
Drug: retifanlimab — retifanlimab will be administered intravenous on Day 1 of each 28 day cycle
  Other Names: INCMGA00012
  Arms: Group B : carboplatin+paclitaxel+retifanlimab

SUMMARY:
This study is a Phase 3 global, multicenter, placebo-controlled double-blind randomized study that will enroll participants with inoperable locally recurrent or metastatic SCAC not previously treated with systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign a written ICF for the study.

  * Are 18 years of age or older (or as applicable per local country requirements).
  * Histologically or cytologically verified, inoperable locally recurrent or metastatic SCAC.
  * No prior systemic therapy other than the following: a. Chemotherapy administered concomitantly with radiotherapy as a radiosensitizing agent is permitted.

    b. Prior neoadjuvant or adjuvant therapy if completed ≥ 6 months before study entry.
  * Has measurable disease per RECIST v1.1 as determined by local site investigator/radiology assessment. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion.
  * Able and willing to provide adequate tissue sample and whole blood sample with central testing result prior to randomization. Biopsy for archival samples should have occurred within 9 months prior to randomization.
  * ECOG performance status 0 to 1.
  * If HIV-positive, then must be stable as defined by: a. CD4+ count ≥ 200/μL, b. Undetectable viral load per standard of care assay, c. Receiving antiretroviral therapy (ART/HAART) for at least 4 weeks prior to study enrollment, and have not experienced any HIV-related opportunistic infection for at least 4 weeks prior to study enrollment.
  * Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Has received prior PD-(L)1 directed therapy
* Has received prior radiotherapy with or without radiosensitizing chemotherapy within 28 days of Cycle 1 Day 1 except for palliative radiation (30 Gy or less) which is restricted for 14 days of Cycle 1 Day 1 (note: all toxicities associated should have resolved to Grade ≤ 1).
* Participants with laboratory outside of the protocol defined ranges.
* History of second malignancy within 3 years (with exceptions).
* Clinically significant pulmonary, cardiac, gastrointestinal or autoimmune disorders.
* Active bacterial, fungal, or viral infections, including hepatitis A, B, and C and IV antibiotic use within 7 days of Cycle 1 Day 1.
* Receipt of a live vaccine within 28 days of planned start of study therapy.
* History of organ transplant, including allogeneic stem cell transplantation.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known hypersensitivity to platinum, paclitaxel, another monoclonal antibody, or any of the excipients that cannot be controlled with standard measures (eg, antihistamines, corticosteroids).
* Participant is pregnant or breastfeeding.
* Current use of protocol defined prohibited medication.
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE v5.
* Inability or unlikely, in the opinion of the investigator, to comply with the Protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (14):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Ochsner Clinic, New Orleans, Louisiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Texas Oncology, Austin, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Renovatio Clinical Consultants Llc, The Woodlands, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Virginia Cancer Specialists, Pc, Arlington, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
- Australia (3):
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre Clayton, Clayton, Victoria
- Belgium (2):
  - Zna Middelheim, Antwerp
  - Ulb Hospital Erasme, Brussels
- Denmark (2):
  - Herlev Og Gentofte Hospital, Herlev
  - Vejle Hospital, Vejle
- France (15):
  - Institut de Cancerologie de L Ouest - Site Paul Papin, Angers
  - Chu Besancon Hospital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Leon Berard, Lyon
  - Chu Hopital de La Timone, Marseille
  - Institut Du Cancer de Montpellier, Montpellier
  - Centre Antoine Laccassagne, Nice
  - Hospital Universitaire Pitie-Salpetriere, Paris
  - Hospital de La Miletrie, Poitiers
  - Chu de Rennes - Hospital Pontchaillou, Rennes
  - Hopital Charles Nicolle Chu Rouen Hospital de Bois-Guillaume, Rouen
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie de Strasbourg, Strasbourg
  - Chu Toulouse Hopital Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitatsklinikum Bonn Aoer, Bonn
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Asklepios Klinik Altona, Hamburg
- Italy (11):
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - European Institute of Oncology, Milan
  - University Di Cagliari-Presidio Policlinico Monserrato, Monserrato
  - Azienda Ospedaliera Universitaria University Degli Studi Della Campania Luigi Vanvitelli, Napoli
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Degli Infermi, Rimini
  - I.R.C.C.S. Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette
- Japan (7):
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Aichi Cancer Center Hospital, Nagoya
  - Osaka International Cancer Institute, Osaka
  - Tohoku University Hospital, Sendai
  - Center Hospital of the National Center For Global Health and Medicine, Shinjuku-ku
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo Universitetssykehus, Oslo
- Panoncology Trials Pan American Center For Oncology Trials, Llc, San Juan, Puerto Rico
- Spain (8):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Son Espases University Hospital, Palma de Mallorca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skaenes Universitetssjukhus Lund, Lund
  - Stockholm South General Hospital Sodersjukhuset, Stockholm
- United Kingdom (12):
  - Royal Sussex County Hospital, Brighton
  - Addenbrooke'S Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - Castle Hill Hospital, Hull
  - Leeds Teaching Hospital, Leeds
  - Royal Free London Nhs Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton
  - Royal Cornwall Hospital Truro Sunrise Centre, Truro

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Rao S, Samalin-Scalzi E, Evesque L, Ben Abdelghani M, Morano F, Roy A, Dahan L, Tamberi S, Dhadda AS, Saunders MP, Casanova N, Guimbaud R, Lievre A, Maurel J, Fakih M, Tian C, Harrison J, Jones MM, Cornfeld M, Spano JP, Rochefort P; POD1UM-303/InterAACT-2 study investigators. Retifanlimab with carboplatin and paclitaxel for locally recurrent or metastatic squamous cell carcinoma of the anal canal (POD1UM-303/InterAACT-2): a global, phase 3 randomised controlled trial. Lancet. 2025 Jun 14;405(10495):2144-2152. doi: 10.1016/S0140-6736(25)00631-2. PMID 40517007
- [Derived] Rao S, Jones M, Bowman J, Tian C, Spano JP. POD1UM-303/InterAACT 2: A phase III, global, randomized, double-blind study of retifanlimab or placebo plus carboplatin-paclitaxel in patients with locally advanced or metastatic squamous cell anal carcinoma. Front Oncol. 2022 Aug 24;12:935383. doi: 10.3389/fonc.2022.935383. eCollection 2022. PMID 36091159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study randomized participants at 70 study centers in Australia, Belgium, Germany, Denmark, Spain, France, the United Kingdom, Italy, Japan, Norway, Puerto Rico, Sweden, and the United States. This report contains data collected through a cutoff date of 15 April 2024.
Groups:
- Retifanlimab 500 mg Q4W + Chemotherapy: Participants received retifanlimab 500 milligrams (mg) every 4 weeks (Q4W) for up to thirteen 28-day cycles (1 year) in the absence of disease progression, intolerable toxicity, death, withdrawal of consent, being lost to follow-up, or premature discontinuation of all assigned study drug administration or for any other reason. Participants also received the standard-of-care chemotherapy regimen of up to 6 induction cycles (24 weeks) of carboplatin (AUC5 on Day 1) and paclitaxel (80 mg per meters squared [mg/m^2] on Days 1, 8, and 15).
- Placebo + Chemotherapy: Participants received matching placebo Q4W for up to thirteen 28-day cycles (1 year) in the absence of disease progression, intolerable toxicity, death, withdrawal of consent, being lost to follow-up, or premature discontinuation of all assigned study drug administration or for any other reason.
- Retifanlimab 500 mg Q4W: In the optional monotherapy treatment period, participants randomized to placebo + chemotherapy who experienced documented progressive disease (PD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) verified by the blinded independent review committee (BICR) had the opportunity to receive open-label retifanlimab monotherapy for up to thirteen 28-day cycles (1 year).
Period: Randomized Period
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Started | 154 | 154 | 0
Received Study Treatment | 154 | 152 | 0
Completed | 0 | 69 (These participants experienced disease progression and transitioned to retifanlimab monotherapy.) | 0
Not Completed | 154 | 85 | 0
Not completed — Ongoing | 90 | 40 | 0
Not completed — Death | 52 | 37 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 0
Not completed — Inclusion Criterion Not Met on Day of Planned Dose | 0 | 1 | 0
Not completed — New Diagnosis of Lymphoma | 1 | 0 | 0
Period: Open-label Monotherapy Period
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Started | 0 | 0 | 69
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 69
Not completed — Ongoing | 0 | 0 | 32
Not completed — Death | 0 | 0 | 35
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.81) | 61.1 (10.51) | 61.3 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 118 | 222
  Male | 50 | 36 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 132 | 137 | 269
  Black/African-American | 3 | 2 | 5
  Asian | 10 | 8 | 18
  Multiple Races | 1 | 0 | 1
  Not Reported | 5 | 3 | 8
  Missing | 0 | 2 | 2
  Mexican | 0 | 1 | 1
  Mixed: White/Indian | 0 | 1 | 1
  White or Other | 1 | 0 | 1
  White British | 1 | 0 | 1
  Captured as "Other" in Database | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 129 | 132 | 261
  Not Reported | 1 | 1 | 2
  Unknown | 10 | 11 | 21
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documented disease progression (PD), according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by blinded independent central review committee (BICR), or death due to any cause, whichever occurred first. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 33.9 months
Population: Full Analysis Set: all randomized participants. Participants were analyzed according to the treatment and strata they had been assigned during randomization. Median PFS time was estimated using the Kaplan-Meier method. The confidence interval for median PFS time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 154 | 154
months | 9.3 [7.5 to 11.3] | 7.4 [7.1 to 7.7]
Statistical Analysis 1: Comparison: Retifanlimab 500 mg Q4W + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p = 0.0006, stratified log-rank test — tested at the 1-sided 2.5% level; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.47 to 0.84] — A stratified Cox regression with Efron's method for tie handling was used to estimate the hazard ratio

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization until the date of death due to any cause.
Time Frame: up to 40.4 months
Reporting Status: Not Posted, anticipated posting 2028-03

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a CR or PR at any post-Baseline visit before the first PD or new anticancer therapy, according to RECIST v1.1 as determined by BICR. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 445 days
Reporting Status: Not Posted, anticipated posting 2028-03

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented response (CR or PR) determined by BICR to the time of first documented disease progression per RECIST v1.1 or death due to any cause. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 32.1 months
Reporting Status: Not Posted, anticipated posting 2028-03

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants maintaining either a confirmed overall response of CR or PR or stable disease (SD) at any post-Baseline visit before the first PD or new anticancer therapy, according to RECIST v1.1 as determined by BICR. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 445 days
Reporting Status: Not Posted, anticipated posting 2028-03

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE ) During the Randomized Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as any AEs either reported for the first time or the worsening of a pre-existing events after the first dose of study treatment and within 90 days of the last administration of retifanlimab/placebo, or within 30 days of the last chemotherapy. AEs that occurred after new anticancer therapy were be excluded.
Time Frame: up to 535 days
Population: Safety Population: all randomized participants who received at least 1 dose of study treatment. Treatment groups for this population were determined according to the actual treatment the participant received regardless of treatment assignment at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 154 | 152
Participants | 154 | 152

7. Secondary Outcome: Number of Participants With Any TEAE Leading to Discontinuation of Study Drug During the Randomized Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as any AEs either reported for the first time or the worsening of a pre-existing events after the first dose of study treatment and within 90 days of the last administration of retifanlimab/placebo, or within 30 days of the last chemotherapy. AEs that occurred after new anticancer therapy were be excluded.
Time Frame: up to 535 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 154 | 152
Participants | 17 | 4

8. Secondary Outcome: Number of Participants With Any TEAE During the Open-label Monotherapy Period
Description: as for outcome 7
Time Frame: up 457 days
Reporting Status: Not Posted, anticipated posting 2028-03

9. Secondary Outcome: Number of Participants With Any TEAE Leading to Discontinuation of Study Drug During the Open-label Monotherapy Period
Description: as for outcome 7
Time Frame: up 457 days
Reporting Status: Not Posted, anticipated posting 2028-03

10. Secondary Outcome: Cmax of Retifanlimab at Steady State When Administered With Carboplatin-paclitaxel
Description: Cmax was defined as the maximum observed plasma concentration of retifanlimab.
Time Frame: preinfusion on Day 1 of Cycles 1, 2, 4, 6, 8, and 12; immediately after infusion on Day 1 of Cycles 1 and 4
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of study treatment and provided at least 1 postdose plasma sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per liter (mg/L)
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Number analyzed (Participants) | 150 | 0 | 0
milligrams per liter (mg/L) | 209 (27.9) |  |

11. Secondary Outcome: Cmin of Retifanlimab at Steady State When Administered With Carboplatin-paclitaxel
Description: Cmin was defined as the minimum observed plasma concentration of retifanlimab.
Time Frame: preinfusion on Day 1 of Cycles 1, 2, 4, 6, 8, and 12; immediately after infusion on Day 1 of Cycles 1 and 4
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Number analyzed (Participants) | 150 | 0 | 0
mg/L | 49.5 (59.4) |  |

12. Secondary Outcome: Tmax of Retifanlimab at Steady State When Administered With Carboplatin-paclitaxel
Description: tmax was defined as the time to the maximum serum concentration of retifanlimab.
Time Frame: preinfusion on Day 1 of Cycles 1, 2, 4, 6, 8, and 12; immediately after infusion on Day 1 of Cycles 1 and 4
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Number analyzed (Participants) | 150 | 0 | 0
hours | 0.720 (35.8) |  |

13. Secondary Outcome: AUC of Retifanlimab at Steady State When Administered With Carboplatin-paclitaxel
Description: AUC was defined as the area under the serum concentration versus time curve.
Time Frame: preinfusion on Day 1 of Cycles 1, 2, 4, 6, 8, and 12; immediately after infusion on Day 1 of Cycles 1 and 4
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day x mg/L
Arm/Group | Retifanlimab 500 mg Q4W + Chemotherapy | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W
Number analyzed (Participants) | 150 | 0 | 0
day x mg/L | 2490 (40.1) |  |

ADVERSE EVENTS:
Time Frame: up to approximately 33 months
Description: Adverse events are reported for all randomized participants who received at least 1 dose of study treatment.
Groups:
- Randomized Period Total: Randomized Period Total
Arm/Group | Placebo + Chemotherapy | Retifanlimab 500 mg Q4W + Chemotherapy | Randomized Period Total | Retifanlimab 500 mg Q4W
All-Cause Mortality (participants affected / at risk) | 38/152 | 53/154 | 91/306 | 35/69
Serious Adverse Events (participants affected / at risk) | 59/152 | 73/154 | 132/306 | 16/69
Other Adverse Events (participants affected / at risk) | 151/152 | 154/154 | 305/306 | 48/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Chemotherapy (N=152) | Retifanlimab 500 mg Q4W + Chemotherapy (N=154) | Randomized Period Total (N=306) | Retifanlimab 500 mg Q4W (N=69)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 5 (5) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 8 (8) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fungating wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Inadequate analgesia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (2) | 5 (6) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 6 (6) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (4) | 0 (0) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 6 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 5 (5) | 9 (9) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urethral fistula (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6) | 2 (2) | 7 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4) | 7 (8) | 0 (0)
Warm autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Chemotherapy (N=152) | Retifanlimab 500 mg Q4W + Chemotherapy (N=154) | Randomized Period Total (N=306) | Retifanlimab 500 mg Q4W (N=69)
Abdominal pain (Gastrointestinal disorders) | 17 (21) | 18 (19) | 35 (40) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 17 (24) | 14 (18) | 31 (42) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (9) | 16 (21) | 23 (30) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 75 (76) | 79 (83) | 154 (159) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 105 (170) | 102 (171) | 207 (341) | 7 (8)
Anxiety (Psychiatric disorders) | 10 (11) | 9 (12) | 19 (23) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (28) | 24 (29) | 45 (57) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 13 (18) | 23 (30) | 5 (6)
Asthenia (General disorders) | 60 (101) | 73 (108) | 133 (209) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (24) | 16 (17) | 36 (41) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 6 (6) | 9 (12) | 15 (18) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 8 (10) | 9 (12) | 3 (3)
COVID-19 (Infections and infestations) | 19 (19) | 20 (21) | 39 (40) | 3 (3)
Constipation (Gastrointestinal disorders) | 61 (85) | 55 (73) | 116 (158) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 17 (22) | 33 (42) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 39 (53) | 37 (44) | 76 (97) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 61 (104) | 74 (158) | 135 (262) | 8 (10)
Dizziness (Nervous system disorders) | 10 (11) | 11 (11) | 21 (22) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (11) | 16 (17) | 1 (1)
Dysgeusia (Nervous system disorders) | 13 (14) | 20 (21) | 33 (35) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 8 (9) | 13 (14) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 23 (25) | 41 (45) | 2 (2)
Dysuria (Renal and urinary disorders) | 5 (5) | 6 (7) | 11 (12) | 4 (5)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9) | 11 (12) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (16) | 21 (23) | 0 (0)
Fatigue (General disorders) | 50 (80) | 45 (56) | 95 (136) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 9 (12) | 12 (15) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 9 (9) | 15 (15) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (4) | 12 (14) | 1 (1)
Headache (Nervous system disorders) | 16 (31) | 25 (29) | 41 (60) | 0 (0)
Hypertension (Vascular disorders) | 11 (17) | 11 (17) | 22 (34) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 12 (12) | 13 (13) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (6) | 10 (11) | 16 (17) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (20) | 19 (24) | 31 (44) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 (19) | 13 (18) | 29 (37) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (8) | 12 (15) | 20 (23) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (5) | 21 (23) | 26 (28) | 8 (8)
Insomnia (Psychiatric disorders) | 10 (12) | 8 (8) | 18 (20) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 17 (29) | 20 (38) | 37 (67) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 9 (14) | 17 (30) | 26 (44) | 1 (1)
Mucosal inflammation (General disorders) | 9 (12) | 17 (18) | 26 (30) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (14) | 22 (25) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 12 (18) | 27 (37) | 1 (1)
Nausea (Gastrointestinal disorders) | 87 (151) | 85 (153) | 172 (304) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 46 (51) | 46 (52) | 92 (103) | 3 (4)
Neurotoxicity (Nervous system disorders) | 13 (13) | 9 (12) | 22 (25) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 67 (199) | 73 (184) | 140 (383) | 2 (2)
Neutrophil count decreased (Investigations) | 34 (72) | 42 (104) | 76 (176) | 0 (0)
Oedema peripheral (General disorders) | 28 (33) | 21 (21) | 49 (54) | 1 (1)
Pain (General disorders) | 6 (7) | 1 (1) | 7 (8) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (12) | 20 (22) | 2 (2)
Paraesthesia (Nervous system disorders) | 18 (23) | 25 (32) | 43 (55) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (15) | 17 (18) | 32 (33) | 0 (0)
Platelet count decreased (Investigations) | 15 (27) | 20 (52) | 35 (79) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 19 (21) | 14 (16) | 33 (37) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 37 (41) | 47 (51) | 4 (5)
Pyrexia (General disorders) | 18 (28) | 21 (36) | 39 (64) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 12 (21) | 24 (29) | 36 (50) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 11 (13) | 17 (21) | 28 (34) | 2 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 9 (9) | 11 (11) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (46) | 22 (38) | 53 (84) | 0 (0)
Urinary tract infection (Infections and infestations) | 18 (25) | 16 (26) | 34 (51) | 3 (4)
Vomiting (Gastrointestinal disorders) | 30 (52) | 37 (50) | 67 (102) | 5 (6)
Weight decreased (Investigations) | 13 (15) | 7 (7) | 20 (22) | 0 (0)
White blood cell count decreased (Investigations) | 20 (50) | 24 (59) | 44 (109) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04472429/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT04472429/SAP_001.pdf